CLINICAL TRIAL: NCT07377045
Title: Phase 1b Dose Escalation Trial of OMTX705, an Anti-Fibroblast Activation Protein Antibody-Drug Conjugate, in Combination With Gemcitabine/Nab-Paclitaxel and Tislelizumab in Patients With Advanced/Metastatic Pancreatic Adenocarcinoma
Brief Title: Clinical Trial of OMTX705 in Combination With Gemcitabine/Nab-Paclitaxel and Tislelizumab in Patients With Advanced/Metastatic Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oncomatryx Biopharma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMTX705-006; 2025-521872-69 (EudraCT Number)
Record Dates: First submitted 2025-12-01; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; tislelizumab

STUDY DESIGN:
Intervention Model Description: The trial consists of two Parts. Part 1 will identify a safe dose of OMTX705 in two novel combinations with gemcitabien/nab-paclitaxel (1A) and with gemcitabine/nab-paclitaxel + tislelizumab (1B). Part 1A and 1B will enroll in a standard 3+3 design.
  Part 2 is a randomized, non-comparative evaluation of preliminary antitumor activity of two combinations of OMTX705: with gemcitabine/nab-paclitaxel and OMTX705+tislelizumab+gemcitabine/nab-paclitaxel vs. a reference arm of gemcitabine/nab-paclitaxel. In part 2, three parallel randomized arms will be opened simultaneously with 1:1:1 randomization (N=15 each).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A (Experimental): Part 1A limited dose escalation arm with three OMTX705 dose levels in combination with gemcitabine/nabpaclitaxel at standard of care doses (starting dose level (DL1A), 4.0 mg/kg; escalating dose level (DL2A) 7.0 mg/kg; reduction dose level (DL-1A 2.0 mg/kg))
  Interventions: Drug: OMTX705; Drug: Nab-paclitaxel + Gemcitabine
- Part 1B (Experimental): Part 1B limited dose escalation arm with three OMTX705 dose levels in combination with gemcitabine/nabpaclitaxel and tislelizumab at standard of care doses (starting dose level (DL1B), 4.0 mg/kg; escalating dose level (DL2B) 7.0 mg/kg; reduction dose level (DL-1B 2.0 mg/kg))
  Interventions: Drug: OMTX705; Drug: Nab-paclitaxel + Gemcitabine; Drug: Tislelizumab (i.v. 200mg)
- Arm 2A (Part 2) (Experimental): OMTX705 at the dose selected by DSMB from Part 1A arm plus gemcitabine/nab-paclitaxel at standard of care doses
  Interventions: Drug: OMTX705; Drug: Nab-paclitaxel + Gemcitabine
- Arm 2B (Part 2) (Experimental): OMTX705 at the dose selected by DSMB from Part 1B arm plus gemcitabine/nab-paclitaxel and tislelizumab at standard of care doses
  Interventions: Drug: OMTX705; Drug: Nab-paclitaxel + Gemcitabine; Drug: Tislelizumab (i.v. 200mg)
- Arm 2C (Part 2) (Other): Reference arm to calibrate safety and efficacy results from the two experimental arms 2A and 2B. Gemcitabine/nab-paclitaxel at standard of care doses.
  Interventions: Drug: Nab-paclitaxel + Gemcitabine

INTERVENTIONS:
Drug: OMTX705 — OMTX705 administered IV at 2.0, 4.0 or 7.5 mg/kg on days 1 and 8 every 21-days cycle
  Arms: Arm 2A (Part 2); Arm 2B (Part 2); Part 1A; Part 1B
Drug: Nab-paclitaxel + Gemcitabine — Gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m2 administered IV on days 1 an8 every 21 days cycle
Drug: Tislelizumab (i.v. 200mg) — Tislelizumab at 200 mg administered IV on day 1 of every 21-days cycle.
  Arms: Arm 2B (Part 2); Part 1B

SUMMARY:
This is a Phase 1b dose escalation trial of OMTX705, an anti-fibroblast activation protein (FAP) antibody-drug conjugate (ADC), in combination with gemcitabine/nab-paclitaxel and tislelizumab in patients with advanced/metastatic pancreatic ductal adenocarcinoma (PDAC).

The trial will be conducted in two parts (Part 1 and Part 2). Both parts will enroll participants with advanced PDAC that, in general, are eligible to receive gemcitabine/nab-paclitaxel. Part 1 is intended to determine the safe recommended dose of OMTX705 in combination with gemcitabine/nab-paclitaxel (1A) and in combination with gemcitabine/nab-paclitaxel+tislelizumab (1B). Both 1A and 1B will enroll in a standard 3+3 design. Only one dose level of OMTX705 will be selected for Part 2 by a Data Safety Monitoring Board (DSMB). In Part 2, 3 parallel randomized arms will be opened simultaneously with 1:1:1 randomization (N=15 each): OMTX705+gemcitabine/nab-paclitaxel (arm 2A), OMTX705+tislelizumab+gemcitabine/nab-paclitaxel (arm 2B) and gemcitabine/nab-paclitaxel (arm 2C, reference arm).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Male and female participant aged 18 years and older.
3. Participants must have histologically or cytologically confirmed PDAC: a) Metastatic PDAC who have not received therapy or received 1 prior line of systemic cytotoxic therapy (Part 1 and Part 2) and if trial treatment is given in the second line setting; b) Non-resectable locoregional PDAC who have not received therapy or received 1 prior line of systemic cytotoxic therapy (Part 1 only); c) A previous treatment with a targeted agent (for example KRAS inhibitor in the context of a clinical trial) without chemotherapy not counted as previous line of therapy. This situation should be discussed with the medical monitor.
4. Participants should have documented disease progression if previously locally advanced disease or be in 2nd line for stage IV or, in the opinion of the investigator, despite of lack of documented PD per image, require a change in the therapy.
5. Participants should be considered in general eligible for standard GA, for first or second line for metastatic disease (Part 1 and 2) or as palliative therapy for non-resectable locoregional cancer (Part 1 only). Patients who received polychemotherapy (FOLFIRINOX or similar) as neoadjuvant/adjuvant treatment and recur locally or distant <6 months after the completion of systemic therapy, will be classified as second line.
6. Measurable disease by RECIST v1.1 on CT PET/CT or magnetic resonance imaging (MRI) scan.
7. Eastern Cooperative Group Performance (ECOG) performance status 0-1.
8. Adequate bone marrow, hepatic and renal function: a) Total bilirubin ≤1.5 times upper limit of normal (ULN) or total bilirubin n <3.0 × ULN with direct bilirubin within normal range in participants with documented Gilbert's syndrome; b) AST and ALT ≤3 times ULN, (if liver metastases are present, then ≤5 times ULN is allowed); c) Serum creatinine ≤1.5 x ULN or creatinine clearance ≥40 mL/min (measured or calculated using the Cockroft-Gault formula); d) Hemoglobin ≥9.0 g/dL (whole or partial blood transfusions not allowed in the two previous weeks); e) ANC ≥1.5 x 109/L (growth factors like granulocyte-colony stimulating factor are not allowed in the two previous weeks); f) Platelet count ≥100 x 109/L (platelet in the two previous weeks transfusions not allowed).
9. Women of childbearing potential (WOCBP) and men with sexual partners who are WOCBP must be willing to adhere to highly effective contraceptive requirements and must agree to avoid impregnating a partner or becoming pregnant, respectively, during the study, and for at least 90 days after the last dose of any IMP. Men with sexual partners who are WOCBP should adhere to contraception requirements for 180 days after the last dose of any IMP.
10. Suitable venous access for safe drug administration and the study-required drug concentration and pharmacodynamics sampling.
11. A valid archival tumor sample.
12. Pretreatment fresh biopsy is optional in Part 1 dose escalation. In Part 2, a fresh pretreatment biopsy and on-treatment is required unless biopsy is associated with significant risk and per discussion with the sponsor medical monitor (or designee).

Exclusion Criteria:

1. Prior treatment with OMTX705 or nab-paclitaxel for the locally advanced (adjuvant or neoadjuvant) for metastatic disease. Previous use of gemcitabine as radiosensitizer or as part of neoadjuvant/adjuvant therapy is allowed if the treatment was completed 6 months before consent signature. Prior treatment with T-cell co-stimulating or immune checkpoint blockade therapies including anti-cytotoxic T-lymphocyte associated protein 4, anti-PD-1, and anti-PD-L1 therapeutic antibodies or any immune checkpoint inhibitor (except for participants to be enrolled in Part 1A).
2. Treatment with systemic anticancer treatments, investigational products, or major surgery within 4 weeks before the first dose of study drug or 5 half-lives, whichever is shorter. Participants should have recovered from previous treatment toxicity to Grade 1, baseline (excluding anemia, lymphopenia, alopecia, and skin pigmentation). Participants with endocrinopathies should have the replacement treatment in stable dosing.
3. History of uncontrolled brain metastasis. Participants with brain metastases are allowed if they are previously treated with surgery, whole-brain radiation, or stereotactic radiosurgery and have brain imaging during screening confirming that brain metastasis are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either MRI or CT and considered controlled with ≤10 mg/day prednisone equivalent at the time of receiving the first dose of OMTX705). For asymptomatic participants, screening brain imaging is not required.
4. Participant has received extended field radiotherapy ≤4 weeks before the start of treatment (≤1 week for limited field radiation for palliation), and who has not recovered to Grade 1 or better from related side effects of such therapy (except for alopecia).
5. Major surgical procedure or significant traumatic injury ≤21 days prior to ICF signature.
6. Cardiac arrhythmias requiring anti-arrhythmic therapy. Note: pacemakers, beta blockers, or digoxin are permitted.
7. Active infection requiring parenteral or oral antibiotics. Antibiotics given for prophylaxis are allowed. They are also allowed for minor localized infections like cystitis, amygdalates or localized skin infections.
8. Evidence of serious uncontrolled medical disorder that, in the opinion of the investigator or medical monitor, makes it unwise for the participant to participate in the study or that might jeopardize compliance with the protocol.
9. Drainage of ascitic or pleural fluid two or more times in the four weeks prior to the first dose of study drug or permanent drain in place (e.g., PleurX®) for ascites or pleural effusion symptom management.
10. Placement of a biliary stent, endoscopic retrograde cholangiopancreatography (ERCP) or biliary catheterization (internal or percutaneous) procedure <7 days before the first dose.
11. Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of AEs or compromised ability to provide written informed consent.
12. Previous or concurrent cancer that is distinct in primary site or histology from PDAC within 3 years prior to randomization except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria]); note: all cancer treatments for cancers that were distinct in a primary site other than PDAC must be completed at least 3 years prior to signature date of the ICF.
13. Uncontrolled or significant cardiovascular disease defined by the New York Hearth Association classification III or IV.
14. History of cerebrovascular stroke or myocardial infarction within the previous 3 months.
15. Grade ≥2 peripheral neuropathy.
16. Received a live vaccine within 30 days prior to first dose of study drug.
17. Known hepatitis B virus surface antigen seropositive or detectable hepatitis C infection viral load. Note: Participants who have positive hepatitis B surface antigen antibody can be included but must have an undetectable hepatitis B viral load. Participants receiving antiviral therapy for hepatitis B virus for any reason are excluded.
18. Participants positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive participants must meet the following criteria: a) have CD4+ T-cell (CD4+) counts ≥350 cells/μL; b) have not had an opportunistic infection within the past 12 months. Participants on prophylactic antimicrobials can be included in the trial; c) should be on established antiretroviral therapy for at least four weeks; d) have an HIV viral load of less than 400 copies/mL prior to enrollment; e) known history of any other relevant congenital or acquired immunodeficiency other than HIV infection.
19. Known or suspected allergy to study treatment or related products, and specifically participants with a prior history of life-threatening reaction to polysorbate 20.
20. Women who are pregnant or breastfeeding or trying to become pregnant.
21. Male participants wishing fathering children, planning for future sperm banking, or expressing concerns about sterility.
22. Participants requiring the concomitant administration of medications that are strong inhibitors or inducers of CYP3A4, 2D6, 1A2, 2C9, 2B6, and 2C19. In case they are taking any of these drugs, they should be stopped at least 14 days prior to first dose.
23. Except Part1A: History of autoimmune disease requiring systemic immunosuppressive therapy (daily prednisone equivalent doses >10 mg/day).
24. Except Part 1A: Participants who discontinued prior treatment with any immune checkpoint due to irAEs, irrespective of grade, recovery, or need for continued steroid therapy. Also, participants without formal contraindication due to previous irAE are not eligible if the AE has not resolved to Grade 1 or better and/or still requires steroids (>10 mg of prednisone equivalent per day) for ongoing management.
25. Except Part 1A: participants with a history of pneumonitis/interstitial lung disease, and participants who discontinued prior immune checkpoint inhibitors due to Grade 2 myocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) during Part 1 of the study | At Day 1, Day 8 and Day 15 of the first 21-day cycle, and up to Day 1 of the second 21-day cycle.
  The nature and frequency of DLTs will be assessed.
Number of participants with treatment emergent adverse events (TEAEs) during Part 1 of the study | From Screening visit through EoT visit (up to 90±5 days after the last dose of study treatment)
  A TEAE is an AE that occurs from the first administration of the study drug up to EoT visit. They can be related to the study drug or not. Frequency, duration, and severity (per CTCAE v.5.0) of TEAEs will be assessed.
Changes in body temperature during Part 1 of the study | At Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  Body temperature should be monitored during each infusion of OMTX705 as follows: on Cycle 1 and 2 before administration and every 30 (±5) minutes thereafter up to 1h ±5 minutes after the end of the infusion (EoI). From Cycle 3 onwards, it will be measured only at OMTX705 pre-dose and in case of clinical symptoms of an infusion-related reaction to document the AE.
Changes in blood pressure (BP) during Part 1 of the study | At Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  BP will be measured in the sitting position after 5 minutes of rest. BP should be monitored during each infusion of OMTX705 as follows: on Cycle 1 and 2 before administration and every 30 (±5) minutes thereafter up to 1h ±5 minutes after the end of the infusion (EoI). From Cycle 3 onwards, it will be measured only at OMTX705 pre-dose and in case of clinical symptoms of an infusion-related reaction to document the AE.
Changes in pulse rate during Part 1 of the study | At Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  Pulse rate will be measured in the sitting position after 5 minutes of rest. Pulse rate should be monitored during each infusion of OMTX705 as follows: on Cycle 1 and 2 before administration and every 30 (±5) minutes thereafter up to 1h ±5 minutes after the end of the infusion (EoI). From Cycle 3 onwards, it will be measured only at OMTX705 pre-dose and in case of clinical symptoms of an infusion-related reaction to document the AE.
Changes in electrocardiogram (ECG) PR interval during Part 1 of the study | At Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in electrocardiogram (ECG) QRS interval during Part 1 of the study | At Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in electrocardiogram (ECG) QT interval during Part 1 of the study | At Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in electrocardiogram (ECG) Fridericia correction QT (QTcF) interval during Part 1 of the study | At Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in concentration of serum chemistry parameters during Part 1 of the study | At Screening visit, at Day 1, Day 8 and Day 15 of the two first 21-day cycles, and at Day 1 and Day 8 of the subsequent 21-day cycles until treatment discontinuation (average of 4 months).
  The following laboratory parameters will be measured for serum chemistry: albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), alkaline phosphatase (ALP), total bilirubin, calcium, creatinine, magnesium, potassium, sodium, lactate dehydrogenase, C-reactive protein, creatine phosphokinase and glucose.
  Chemistry C1D1 blood samples may be collected within 3 days before dosing to ensure participant eligibility. If screening clinical laboratory testing was performed within 3 days before the C1D1 dose, it does not need to be repeated. Chemistry blood samples will be obtained weekly for the first 2 cycles (Day 1, 8 and 15 of Cycle 1 and Cycle 2). From Cycle 3, chemistry will be collected only on the administration days (Day 1 and Day 8). Samples can be collected and analyzed the day before.
Changes in concentration of hematology parameters during Part 1 of the study | At Screening visit, at Day 1, Day 8 and Day 15 of the two first 21-day cycles, and at Day 1 and Day 8 of the subsequent 21-day cycles until treatment discontinuation (average of 4 months).
  The following laboratory parameters will be measured for hematology: hemoglobin, platelet count, red blood cell count , white blood cells (WBC) count and differential WBC count (absolute number).
  Hematology C1D1 blood samples may be collected within 3 days before dosing to ensure participant eligibility. If screening clinical laboratory testing was performed within 3 days before the C1D1 dose, it does not need to be repeated. Hematology blood samples will be obtained weekly for the first 2 cycles (Day 1, 8 and 15 of Cycle 1 and Cycle 2). From Cycle 3, hematology will be collected only on the administration days (Day 1 and Day 8). Samples can be collected and analyzed the day before.
Treatment modifications during Part 1 of the study | From Screening visit and through the study until treatment discontinuation (average of 4 months).
  Treatment modifications are measured as percentage of relative dose intensity.
Definition of Maximum tolerated dose (MTD) for Part 2 | From Screening visit and through the study until treatment discontinuation (average of 4 months).
  MTD definition for Part 2: recommended dose will be based on MTD, or in absence of MTD based on non-DLT safety, efficacy as well as other relevant pharmacokinetics/pharmacodynamics evaluations.
Objective response rate (ORR) during Part 2 of the study | From Screening visit through EoT1 visit (30 ±2 days after the last dose of study treatment)
  The ORR is defined as the proportion of participants who have a confirmed partial response (PR) or complete response (CR) to study treatment per RECIST v1.1 as determined by the investigator.

SECONDARY OUTCOMES:
Disease control rate (DCR) | From Screening visit through EoT1 visit (30 ±2 days after the last dose of study treatment).
  DCR was assessed according to RECIST 1.1 criteria and defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD).
Duration of response (DoR) | From Screening visit through EoT1 visit (30 ±2 days after the last dose of study treatment).
  DoR following following RECIST 1.1 criteria.
Time to response | From Screening visit through EoT1 visit (30 ±2 days after the last dose of study treatment)
  Time to response following RECIST 1.1 criteria.
Progression-free survival (PFS) | From Screening visit through the study until last PFS-FU visit (average of 4 months)
  Time from enrollment to disease progression or death, whichever occurred first, assessed according to RECIST 1.1 criteria.
  Participants who discontinue study treatment for reasons other than progression disease (PD) will continue to attend progression-free survival follow-up (PFS-FU) visits every 12 (±1) weeks from the EoT1 visit until the occurrence of PD, loss to folow-up, consent withdrawal, death, the start of subsequent systemic antineoplastic therapy, or study termination, whichever occurs first.
Proportion of participants without progression/death | At 3, 6 and 12 months
  Percentage of participants who remained alive and free of disease progression according to RECIST 1.1 criteria at each timepoint
Overall survival (OS) | From Screening visit through the study until last OS-FU visit (average of 4 months)
  OS is defined as the time from enrollment to death from any cause. Participants' survival information (alive/dead and date of death) will be assessed every 3 months from the first dose of OMTX705 through participant contact (by phone or hospital visit) or at the time the death becomes known. If the site is aware that a patient is deceased, the date of death should be recorded in the eCRF without waiting for the next OS visit.
Proportion of participants alive | At 3, 6, 12 and 18 months
  Percentage of participants alive at each timepoint
Percentage of reduction in cancer antigen 19-9 (CA19-9) from baseline upon treatment | Part 1 and 2 (Arm 2A/2B): Screening and Day 1 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Part 2 (Arm 2C): Screening and Day 1 of each 28-day cycle until treatment discontinuation (average of 4 months).
  Changes in CA19-9 concentration from baseline upon treatment. CA19-9 will be measured locally in all participants at Screening and Day 1 of every cycle.
Quantification (titer) of anti-drug antibodies (ADAs) against OMTX705 | Part 1 and 2 (Arm 2A/2B): At Day 1 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  The formation of ADAs against OMTX705 will be assessed in blood samples collected prior to OMTX705 administration at Day 1 of each cycle, EoT1 and PFS-FU. The ADAs will be measured in a central laboratory designated by the sponsor. ADAs will not be assessed in Arm 2C.
Percentage of ADA-positive participants | Part 1 and 2 (Arm 2A/2B): At Day 1 of each 21-day cycle through the study until treatment discontinuation (average of 4 months).
  Percentage of participants who develop detectable ADAs to OMTX705. The formation of ADAs against OMTX705 will be assessed in blood samples collected prior to OMTX705 administration at Day 1 of each cycle, EoT1 and PFS-FU. The ADAs will be measured in a central laboratory designated by the sponsor. ADAs will not be assessed in Arm 2C.
Blood concentrations of conjugated antibody | Part 1 and 2 (Arm 2A/2B): At Day 1, Day 8 and Day 15 of Cycle 1, and at Day 1 and Day 8 of Cycle 2 and Cycle 4 (each cycle is 21 days).
  Blood concentrations of conjugated antibody will be listed and summarized using descriptive statistics. The measurement of conjugated antibody will be performed using validated methods at a central laboratory designated by the sponsor.
  Plasma/serum samples will be collected in Cycle 1, Cycle 2 and Cycle 4 on: Day 1 (predose, end of infusion, 1-2 hours post-infusion and 2-4 hours post-infusion), on Day 8 (predose and end of infusion), and on Day 15 (±24 hours, cycle 1 only). No collection will be performed in Arm 2C.
Blood concentrations of unconjugated payload (TAM470) | Part 1 and 2 (Arm 2A/2B): At Day 1, Day 8 and Day 15 of Cycle 1, and at Day 1 and Day 8 of Cycle 2 and Cycle 4 (each cycle is 21 days).
  Blood concentrations of TAM470 will be listed and summarized using descriptive statistics. The measurement of TAM470 will be performed using validated methods at a central laboratory designated by the sponsor.
  Plasma/serum samples will be collected in Cycle 1, Cycle 2 and Cycle 4 on: Day 1 (predose, end of infusion, 1-2 hours post-infusion and 2-4 hours post-infusion), on Day 8 (predose and end of infusion), and on Day 15 (±24 hours, cycle 1 only). No collection will be performed in Arm 2C.
Number of participants with dose limiting toxicities (DLTs) during Part 2 of the study | Arm 2A/2C: At Day 1, Day 8 and Day 15 of the first 21-day cycle, and up to Day 1 of the second 21-day cycle. Arm 2C: At Day 1, Day 8 and Day 15 of the first 28-day cycle, and up to Day 1 of the second 28-day cycle.
  The nature and frequency of DLTs will be assessed.
Number of participants with treatment emergent adverse events (TEAEs) during Part 2 of the study | From Screening visit through EoT visit (up to 90±5 days after the last dose of study treatment)
  A TEAE is an AE that occurs from the first administration of the study drug up to EoT visit. They can be related to the study drug or not. Frequency, duration, and severity (per CTCAE v.5.0) of TEAEs will be assessed.
Changes in body temperature during Part 2 of the study | Arm 2A/2B: Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Arm 2C: Screening visit, Day 1 and Day 8 of each 28-day cycle until treatment discontinuation (average of 4 months).
  Body temperature should be monitored during each infusion of OMTX705 as follows: on Cycle 1 and 2 before administration and every 30 (±5) minutes thereafter up to 1h ±5 minutes after the end of the infusion (EoI). From Cycle 3 onwards, it will be measured only at OMTX705 pre-dose and in case of clinical symptoms of an infusion-related reaction to document the AE.
Changes in blood pressure (BP) during Part 2 of the study | Arm 2A/2B: Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Arm 2C: Screening visit, Day 1 and Day 8 of each 28-day cycle until treatment discontinuation (average of 4 months).
  BP will be measured in the sitting position after 5 minutes of rest. BP should be monitored during each infusion of OMTX705 as follows: on Cycle 1 and 2 before administration and every 30 (±5) minutes thereafter up to 1h ±5 minutes after the end of the infusion (EoI). From Cycle 3 onwards, it will be measured only at OMTX705 pre-dose and in case of clinical symptoms of an infusion-related reaction to document the AE.
Changes in pulse rate during Part 2 of the study | Arm 2A/2B: Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Arm 2C: Screening visit, Day 1 and Day 8 of each 28-day cycle until treatment discontinuation (average of 4 months).
  Pulse rate will be measured in the sitting position after 5 minutes of rest. Pulse rate should be monitored during each infusion of OMTX705 as follows: on Cycle 1 and 2 before administration and every 30 (±5) minutes thereafter up to 1h ±5 minutes after the end of the infusion (EoI). From Cycle 3 onwards, it will be measured only at OMTX705 pre-dose and in case of clinical symptoms of an infusion-related reaction to document the AE.
Changes in electrocardiogram (ECG) PR interval during Part 2 of the study | Arm 2A/2B: Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Arm 2C: Screening visit, Day 1 and Day 8 of each 28-day cycle until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in electrocardiogram (ECG) QRS interval during Part 2 of the study | Arm 2A/2B: Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Arm 2C: Screening visit, Day 1 and Day 8 of each 28-day cycle until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in electrocardiogram (ECG) QT interval during Part 2 of the study | Arm 2A/2B: Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Arm 2C: Screening visit, Day 1 and Day 8 of each 28-day cycle until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in electrocardiogram (ECG) Fridericia correction QT (QTcF) interval during Part 2 of the study | Arm 2A/2B: Screening visit, Day 1 and Day 8 of each 21-day cycle through the study until treatment discontinuation (average of 4 months). Arm 2C: Screening visit, Day 1 and Day 8 of each 28-day cycle until treatment discontinuation (average of 4 months).
  Changes in ECG assessed using a 12-lead ECG machine. In Cycle 1 and Cycle 2 ECGs will be recorded before the start of OMTX705 infusion and after the end of infusion (+15 minutes).
Changes in concentration of serum chemistry parameters during Part 2 of the study | At Screening visit, at Day 1, Day 8 and Day 15 of Cycle 1 and Cycle 2, and at Day 1 and Day 8 of subsequent cycles through the study until treatment discontinuation (average of 4 months) (Arm 2A/2B: each cycle is 21 days; Arm 2C: each cycle is 28 days).
  The following laboratory parameters will be measured for serum chemistry: albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), alkaline phosphatase (ALP), total bilirubin, calcium, creatinine, magnesium, potassium, sodium, lactate dehydrogenase, C-reactive protein, creatine phosphokinase and glucose.
  Chemistry C1D1 blood samples may be collected within 3 days before dosing to ensure participant eligibility. If screening clinical laboratory testing was performed within 3 days before the C1D1 dose, it does not need to be repeated. Chemistry blood samples will be obtained weekly for the first 2 cycles (Day 1, 8 and 15 of Cycle 1 and Cycle 2). From Cycle 3, chemistry will be collected only on the administration days (Day 1 and Day 8). Samples can be collected and analyzed the day before.
Changes in concentration of hematology parameters during Part 2 of the study | At Screening visit, at Day 1, Day 8 and Day 15 of Cycle 1 and Cycle 2, and at Day 1 and Day 8 of subsequent cycles through the study until treatment discontinuation (average of 4 months) (Arm 2A/2B: each cycle is 21 days; Arm 2C: each cycle is 28 days).
  The following laboratory parameters will be measured for hematology: hemoglobin, platelet count, red blood cell count , white blood cells (WBC) count and differential WBC count (absolute number).
  Hematology C1D1 blood samples may be collected within 3 days before dosing to ensure participant eligibility. If screening clinical laboratory testing was performed within 3 days before the C1D1 dose, it does not need to be repeated. Hematology blood samples will be obtained weekly for the first 2 cycles (Day 1, 8 and 15 of Cycle 1 and Cycle 2). From Cycle 3, hematology will be collected only on the administration days (Day 1 and Day 8). Samples can be collected and analyzed the day before.
Treatment modifications during Part 2 of the study | From Screening visit and through the study until treatment discontinuation (average of 4 months).
  Treatment modifications are measured as percentage of relative dose intensity.

CONTACTS AND LOCATIONS:
Locations (7):
- Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts, United States
- Spain (6):
  - Hospital Universitario Vall d'Hebron (VHIO), Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - ICO- Hospitalet Catalan Institute of Oncology, L'Hospitalet de Llobregat
  - Hospital Universitario 12 Octubre, Madrid
  - Clinica Universidad de Navarra (CUN), Pamplona
  - Hospital Clínico Universitario de Santiago - CHUS, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No